CLINICAL TRIAL: NCT00056927
Title: Preventing Initiation of Smoking by Children
Brief Title: Anti-Smoking Program for Parents: Effects on Child Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: 2R01HD36514-5; 2R01HD036514 (NIH)
Record Dates: First submitted 2003-03-26; First posted 2003-03-27 (Estimated); Last update posted 2006-10-02 (Estimated); Status verified 2005-07

CONDITIONS: Smoking
Keywords: Smoking; Primary Prevention; Health Education; Child; Parents; Parenting Education; Communication
MeSH Terms: conditions — Smoking; Health Education; Communication

INTERVENTIONS:
Behavioral: Anti-smoking Socialization Program

SUMMARY:
The purpose of this study is to determine whether an anti-smoking program for parents who smoke will lower the odds that their children will start smoking. The study will evaluate an activity-based program for parents and their children. The program is home-based and uses the mail for program delivery.

DETAILED DESCRIPTION:
Youth whose parents smoke cigarettes are at high risk for early initiation of cigarette smoking, and youth who first smoke cigarettes during childhood are at high risk for subsequent addiction to tobacco. Parents influence their children's perceptions of the prevalence of smoking, the acceptability of smoking, the accessibility of cigarettes, and the personal and social consequences of smoking. All parents, including parents who smoke, can engage in anti-smoking socialization, which may lower children's risk of smoking.

Although there are some programs available that are directed at preventing initiation of smoking during childhood, none of these prevention programs engage parents who smoke in altering children's smoking-specific socialization. This study will evaluate a program to change smoking-specific socialization of children in households where parents smoke cigarettes.

Consenting volunteers will be randomly assigned to either treatment (anti-smoking socialization program) or control groups. Parents in the treatment group will participate in the "Smoke-free Kids" program and receive activity magazines, newsletters, and support calls. Parents in the control group will receive a fact sheet about youth smoking. Parents involved in the study will be assessed through a telephone interview 1 month after completion of the three-month anti-smoking program. Assenting children will complete surveys administered at school at 12, 24, and 36 months after completion of the anti-smoking program. Primary and secondary dependent variables include initiation of cigarette smoking and susceptibility to cigarette smoking by children. The child survey will also assess risk and protective factors.

ELIGIBILITY:
Inclusion Criteria

* Parents or guardians who smoke
* Have children in the 3rd grade
* Belong to participating school districts in North Carolina, South Carolina, or Colorado

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1007
Dates: Start 1997-09; Study Completion 2002-08

PRIMARY OUTCOMES:
Initiation of cigarette smoking -- 3 years post treatment

SECONDARY OUTCOMES:
Susceptibility for initiation of cigarette smoking -- 1 year post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Jackson, Ph.D., Principal Investigator — Pacific Institute for Research and Evaluation

REFERENCES:
- [Background] Jackson C, Dickinson D. Can parents who smoke socialise their children against smoking? Results from the Smoke-free Kids intervention trial. Tob Control. 2003 Mar;12(1):52-9. doi: 10.1136/tc.12.1.52. PMID 12612363